CLINICAL TRIAL: NCT05445063
Title: Safety and Efficacy of Autologous Transplantation of Induced Pluripotent Stem Cell-Derived Retinal Pigment Epithelium in the Treatment of Macular Degeneration
Brief Title: Safety and Efficacy of Autologous Transplantation of iPSC-RPE in the Treatment of Macular Degeneration
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-214
Record Dates: First submitted 2022-06-05; First posted 2022-07-06 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-03

CONDITIONS: Macular Degeneration
Keywords: Retinal disease; Macular degeneration; Stem Cells; RPE; Safety; Efficacy
MeSH Terms: conditions — Macular Degeneration; Retinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants receiving intervention (Experimental): Participants will receive autologous transplantation of induced pluripotent stem cell-derived retinal pigment epitheliums.
  Interventions: Biological: Autologous iPSC-derived RPE

INTERVENTIONS:
Biological: Autologous iPSC-derived RPE — Autologous transplantation of iPSC-derived RPE

SUMMARY:
This project intends to perform autologous transplantation of induced pluripotent stem cell-derived retinal pigment epithelium (iPSC-RPE). The clinical-grade RPE will be transplanted into subretinal space to treat refractory age-related macular degeneration. The efficacy and safety of RPE transplants to treat macular degeneration will be monitored and analyzed with results from EDTRS, BCVA, OCT, ERG, microperimetry, and fluorescein angiography, before and after the treatment.

DETAILED DESCRIPTION:
The investigators will generate iPSC lines from recruited participants and differentiate the iPSC into RPE. Autologous iPSC-derived RPE will be transplanted into participants eyes by subretinal injections. The safety and efficacy will be closely monitored and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50-75 years;
* Clinical diagnosis is consistent with the definition of late dry AMD in the age-related eye disease study (AREDS), with one or more >250 um geographic atrophy in the fovea;
* Clinical diagnosis is wet AMD, but no obvious efficacy after conventional treatment;
* The BCVA of the target eye will be 0.05 to 0.3;
* Voluntary as test subjects, informed consent, regular follow-up on time.

Exclusion Criteria:

* One-eyed subjects;
* Macular atrophy caused by other diseases in addition to AMD;
* Suffer from retinitis pigmentosa, choroidal retinitis, central serous choroiditis, diabetic retinopathy, or other retinal vascular and degenerative diseases besides AMD;
* Lens opacities (affecting the central vision), glaucoma, uveitis, retinal detachment, optic neuropathy, and other ocular histories;
* Other intraocular surgery histories besides cataract surgery;
* Combined with severe systemic diseases, such as heart failure, liver disease, renal insufficiency, cor pulmonale, COPD in the previous 12 months;
* Combined with severe infectious diseases, such as HIV, HBV, HCV, syphilis, tuberculosis, etc;
* Abnormal blood coagulation function or other laboratory tests;
* If female and of childbearing potential, pregnant, breastfeeding, or planning to become pregnant through the study;
* If male, refuse to use barrier and spermicide contraception during the study;
* Malignant tumor and history of malignancy;
* Any immune deficiency;
* Allergy to tacrolimus or other macrolides;
* Any immune deficiency;
* Use glucocorticoids, immunosuppressive drugs, or antipsychotic drugs in the previous 3 months;
* Use anticoagulant, or the platelet function is still not restored to normal after stopping antiplatelet drugs for 10 days;
* A history of addiction to alcoholism or prohibited drugs;
* Be participating in other intervention clinical trials or receiving other study medications;
* Poor compliance, difficulty to complete the study, or refusal to informed consent;
* Some other situations which might increase the risks of the subjects or interfere with clinical trials, such as mental disorders, cognitive dysfunction, etc.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Safety measure | 12 months
  Safety will be assessed by Adverse Events (AEs) of special interest in regards to the investigational product. This will include obtaining information about Serious Adverse Events (SAEs) that are neurologic, infectious, hematologic or fatal, any AE that causes the subject to withdraw from the study, any new diagnosis of an ocular or immune-mediated disorder, cancer (irrespective of prior history), ectopic or proliferative cell growth (RPE or non-RPE) with adverse clinical consequence, unexpected, clinically significant AE possibly related to the cell transplant procedure or the investigational product (autologous iPSC-RPE), pregnancy in a female subject or the partner of a male subject and pregnancy outcome.

SECONDARY OUTCOMES:
Best Corrected Visual Acuity (BCVA) | 12 months
  Change in visual acuity will be measured by Early Treatment Diabetic Retinopathy Study (ETDRS) chart.
Optical coherence tomography (OCT) imaging | 12 months
  The number of patients with serious retinal detachment, retinal hemorrhage, and cystoid macular edema, and the change in target treatment areas.
Color and autofluorescence imaging | 12 months
  Change in target treatment areas.
Fluorescein angiography | 12 months
  Change in target treatment areas.
Fundus autofluorescence | 12 months
  Change in target treatment areas.
Microperimetry | 12 months
  Exploratory evaluations for the change of retinal sensitivity from baseline in the region of interest.
Electroretinography (ERG) | 12 months
  Exploratory evaluations for the change of retinal electrophysiology responses from baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tongren Hospitol,Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Detailed plan will be made based on institute regulations and funder policies. The investigators will adjust the plan case-by-case accordingly.